CLINICAL TRIAL: NCT05499390
Title: A Randomized Controlled, Multi-center Phase III Clinical Trial of AK112 Versus Pembrolizumab as First-line Treatment for PD-L1-Positive Locally-Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: AK112 in Advanced Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK112-303
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Advanced Non-small-cell Lung Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK112 (Experimental): Subjects receive AK112 monotherapy intravenously (IV), selected dose.
  Interventions: Drug: AK112
- Pembrolizumab (Active Comparator): Subjects receive Pembrolizumab monotherapy intravenously (IV), 200mg q3w.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: AK112 — Subjects receive AK112 intravenously.
  Arms: AK112
Drug: Pembrolizumab — Subjects receive Pembrolizumab intravenously.
  Arms: Pembrolizumab

SUMMARY:
This trial is a Phase III study. All patients are stage IIIB/C (unsuitable for radical therapy) or IV non-small cell lung cancer(NSCLC), Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The purpose of this study is to evaluate the efficacy and safety of AK112 comparing Pembrolizumab in subjects with advanced NSCLC whose tumors have a programmed cell death-ligand 1 (PD-L1) Tumor Proportion Score (TPS) greater than or equal to 1%.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of NSCLC.
* Has Stage IIIB/C or IV NSCLC (American Joint Committee on Cancer [AJCC]).
* ≥18 years old (at the time consent is obtained).
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue.
* Has a life expectancy of at least 3 months.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the site study team.
* Has no EGFR-sensitive mutations or ALK gene translocations.
* Has positive PD-L1 expression in tumor tissue.
* Has no prior systemic anti-tumor therapy for locally advanced or metastatic NSCLC.
* Has adequate organ function.
* Has recovered from the effects of any prior radiotherapy or surgery.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Has any histologically small cell carcinoma component.
* Is currently participating in a study of an investigational agent or using an investigational device.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy within 2 years prior to the first dose of study treatment.
* Has undergone major surgery within 30 days of Study Day 1.
* Has a known additional malignancy that is progressing or requires systemic treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has an active infection requiring systemic therapy.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* History of myocardial infarction, unstable angina, congestive heart failure within 12 months prior to day 1 of study treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy.
* Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment.
* Has any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by IRRC per RECIST v1.1 | Up to 2 approximately years
  Progression-free survival (PFS) is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the blinded IRRC or death due to any cause (whichever occurs first).

SECONDARY OUTCOMES:
OS | Up to 2 approximately years
  Overall Survival (OS) is defined as the time from the start of treatment with AK112 until death due to any cause.
ORR assessed by IRRC per RECIST v1.1 | Up to 2 approximately years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1.
DoR assessed by IRRC per RECIST v1.1 | Up to 2 approximately years
  Duration of response (DoR) assessed according to RECIST v1.1.
DCR assessed by IRRC per RECIST v1.1 | Up to 2 approximately years
  Disease control rate (DCR) assessed according to RECIST v1.1.
TTR assessed by IRRC per RECIST v1.1 | Up to 2 approximately years
  Time to response (TTR) is defined as the time to response base on RECIST v1.1.
PFS assessed by investigator per RECIST v1.1 | Up to 2 approximately years
  Progression-free survival (PFS) is defined as the time from the date of randomization till the first documentation of disease progression assessed by the investigator or death due to any cause (whichever occurs first).
ORR assessed by the investigator per RECIST v1.1 | Up to 2 approximately years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1.
DoR assessed by the investigator per RECIST v1.1 | Up to 2 approximately years
  Duration of response (DoR) assessed according to RECIST v1.1.
DCR assessed by the investigator per RECIST v1.1 | Up to 2 approximately years
  Disease control rate (DCR) assessed according to RECIST v1.1.
TTR assessed by the investigator per RECIST v1.1 | Up to 2 approximately years
  Time to response (TTR) is defined as the time to response base on RECIST v1.1.
AE | Up to 2 approximately years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
ADA | Up to 2 approximately years
  Number of subjects with detectable anti-drug antibodies (ADA).
PD-L1 expression | Up to 2 approximately years
  The correlationship between PD-L1 expression and AK112 anti-tumor activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang L, Yao W, Shen H, Xie C, Chen H, Chen K, Su W, Gan X, Zhuo M, Chen E, Xu Z, Zhang Y, Wang M, Ma R, Wu H, Zhang Z, Ye F, Moore AC, Zhou C. Plain language summary: comparing ivonescimab with pembrolizumab in people with PD-L1-positive non-small cell lung cancer in the HARMONi-2 study. Future Oncol. 2026 Jan;22(1):27-36. doi: 10.1080/14796694.2025.2601138. Epub 2025 Dec 28. PMID 41457351
- [Derived] Xiong A, Wang L, Chen J, Wu L, Liu B, Yao J, Zhong H, Li J, Cheng Y, Sun Y, Ge H, Yao J, Shi Q, Zhou M, Chen B, Han Z, Wang J, Bu Q, Zhao Y, Chen J, Nie L, Li G, Li X, Yu X, Ji Y, Sun D, Ai X, Chu Q, Lin Y, Hao J, Huang D, Zhou C, Shan J, Yang H, Liu X, Wang J, Shang Y, Mei X, Yang J, Lu D, Hu M, Wang ZM, Li B, Xia M, Zhou C. Ivonescimab versus pembrolizumab for PD-L1-positive non-small cell lung cancer (HARMONi-2): a randomised, double-blind, phase 3 study in China. Lancet. 2025 Mar 8;405(10481):839-849. doi: 10.1016/S0140-6736(24)02722-3. PMID 40057343